CLINICAL TRIAL: NCT05715671
Title: Effect of Subanesthetic Dose of Esketamine on Sleep Quality and Recovery of Gastrointestinal Function in Patients Undergoing General Anesthesia Laparoscopic Uterine Surgery in the Early Postoperative Period
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zhuan Zhang (Other)
Responsible Party: Sponsor-Investigator, Zhuan Zhang, Clinical Professor, Yangzhou University
Organization: Yangzhou University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 20221217
Record Dates: First submitted 2022-12-17; First posted 2023-02-08 (Actual); Last update posted 2024-05-21 (Actual); Status verified 2024-05

CONDITIONS: Patients Undergoing General Anesthesia Laparoscopic Uterine Surgery
Keywords: Esketamine; General anesthesia laparoscopic uterine surgery; Sleep quality; Recovery of gastrointestinal function
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Esketamine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Esketamine for induction 0.15mg/kg and maintenance 0.15mg/kg/h (Experimental)
  Interventions: Drug: esketamine
- Esketamine for induction 0.3mg/kg and maintenance 0.3mg/kg/h (Experimental)
  Interventions: Drug: esketamine
- No esketamine (No Intervention)

INTERVENTIONS:
Drug: esketamine — The corresponding esketamine dose for each group was used at the end of anesthesia induction, and esketamine was changed to the corresponding maintenance dose for each group prior to surgical skin incision.
  Arms: Esketamine for induction 0.15mg/kg and maintenance 0.15mg/kg/h; Esketamine for induction 0.3mg/kg and maintenance 0.3mg/kg/h

SUMMARY:
Patients undergoing gynecological surgery are at high risk of developing postoperative sleep disorders. Intraoperative opioid use is detrimental to the patient's postoperative recovery of gastrointestinal function. Esketamine has sedative, hypnotic, analgesic, inflammatory response suppression, and antidepressant effects. Its hypnotic mechanism may be related to its rapid blockade of NMDA receptors and hyperpolarization-activated cyclic nucleotide-gated cation channels. Also can reduce the application of perioperative opioids, which in turn promotes the recovery of gastrointestinal function in patients after surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 40 and 65 years;
2. ASA class I-III;
3. Proposed laparoscopic total hysterectomy/myomectomy;
4. Operative time ≥ 1 h;
5. Body mass index of 18-30 kg/m2.

Exclusion Criteria:

1. Patient refusal;
2. Known allergy to anesthetic drugs;
3. Preoperative sleep disorder (Pittsburgh Sleep Quality Index [PSQI] > 7);
4. Severe hypertension, coronary artery disease, cardiac insufficiency, pulmonary hypertension, pulmonary heart disease, increased cranial pressure, increased intraocular pressure, seizures, shift work, obstructive sleep apnea syndrome;
5. Long-term use of opioids or sedative-hypnotic drugs;
6. History of psychiatric or neurological disease;
7. Previous or planned neurosurgery.

(7)hearing or visual impairment that precludes a scale assessment.

Ages: 40 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Actual)
Dates: Start 2023-03-25 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Changes in the level of actigraphy | Baseline (the night before surgery), postoperative nights 1 and 2
  Through the actigraphy, monitor the patient's sleep quality.
Changes in the level of Pittsburgh sleep quality index | Baseline (the night before surgery), postoperative nights 1, 2 and 3
  Assess the patient's sleep quality by asking questions on the scale on a scale of 0-21, with higher scores representing poorer sleep quality.

SECONDARY OUTCOMES:
Changes in the level of Mean Arterial Pressure | Baseline (before induction), after loading dose of intervention, at the beginning of surgery, upon surgery completion, immediately after extubation, and 30min after transfer to the post-anesthesia care unit
  The outcome above should be measured at the time before induction, after loading dose of intervention, at the beginning of surgery, upon surgery completion, immediately after extubation, and 30min after transfer to the post-anesthesia care unit.
Changes in the level of IL-6 | Preoperatively, upon surgery completion, postoperative day 1
  The above results should be measured preoperatively, upon surgery completion, and on the 1st postoperative day.
Changes in the level of Melatonin | Preoperatively, upon surgery completion, postoperative day 1
  The above results should be measured preoperatively, upon surgery completion, and on the 1st postoperative day.
Changes in the level of BDNF | Preoperatively, upon surgery completion, postoperative day 1
  The above results should be measured preoperatively, upon surgery completion, and on the 1st postoperative day.
Changes in the level of IL-10 | Preoperatively, upon surgery completion, postoperative day 1
  The above results should be measured preoperatively, upon surgery completion, and on the 1st postoperative day.
Changes in the level of Heart Rate | Baseline (before induction), after loading dose of intervention, at the beginning of surgery, upon surgery completion, immediately after extubation, and 30min after transfer to the post-anesthesia care unit
  The outcome above should be measured at the time before induction, after loading dose of intervention, at the beginning of surgery, upon surgery completion, immediately after extubation, and 30min after transfer to the post-anesthesia care unit.
Changes in the level of Oxygen saturation | Baseline (before induction), after loading dose of intervention, at the beginning of surgery, upon surgery completion, immediately after extubation, and 30min after transfer to the post-anesthesia care unit
  The outcome above should be measured at the time before induction, after loading dose of intervention, at the beginning of surgery, upon surgery completion, immediately after extubation, and 30min after transfer to the post-anesthesia care unit.
Changes in the level of the visual analogue scale | Postoperative days 1 and 2
  Assess the patient's pain by asking on a scale of 0-10, with higher scores representing more severe pain.
Recovery of gastrointestinal function | Postoperative first 1 day
  Record the time of the first postoperative exhausting
Recovery of gastrointestinal function | Postoperative first 1 day
  Record the time of the first postoperative bowel movement
Recovery of gastrointestinal function | Postoperative first 1 day
  Record the time of the first postoperative feeding
Postoperative adverse reactions | Postoperative day 1
  Record the occurrence of adverse reactions (nausea and vomiting, nightmares, dizziness, and mirages) on the 1st postoperative day.

CONTACTS AND LOCATIONS:
Overall Officials: zhuan zhang, professor, Principal Investigator — The Affiliated Hospital of Yangzhou University
Locations (1):
- the Affiliated Hospital of Yangzhou University, Yangzhou, Jiangsu, China

REFERENCES:
- [Derived] Yuan B, Tian S, Pu X, Yin J, Wang M, Feng S, Lv X, Sun Y, Yao H, Li M, Li S, Zhang Z. Esketamine improves postoperative sleep quality in women undergoing gynecological laparoscopy: A prospective, randomized, double-blind, and controlled trial. Sleep Med. 2025 Dec;136:106852. doi: 10.1016/j.sleep.2025.106852. Epub 2025 Oct 14. PMID 41115350